CLINICAL TRIAL: NCT06109662
Title: Multimorbidity and Sarcopenia Feasibility Study in Chronic Kidney Disease
Acronym: MaSS-CKD
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 328554
Record Dates: First submitted 2023-10-13; First posted 2023-10-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Sarcopenia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy volunteers: Normal renal function with no kidney disease. Participants with other comorbidities can be included as long as not listed on the exclusion criteria. They will have body composition measured, and eGFR measured.
  Interventions: Diagnostic Test: Cystatin C eGFR; Other: Bioimpedance Analysis (Body composition analysis)
- Chronic Kidney Disease Stage 3: People with CKD Stage 3 (eGFR 30-59). They will have body composition measured, and eGFR measured.
  Interventions: Diagnostic Test: Cystatin C eGFR; Other: Bioimpedance Analysis (Body composition analysis)
- Chronic Kidney Disease Stage 4: People with CKD 4 (eGFR 15-29). They will have body composition measured, and eGFR measured.
  Interventions: Diagnostic Test: Cystatin C eGFR; Other: Bioimpedance Analysis (Body composition analysis)
- Chronic Kidney Disease Stage 5: People with CKD 5 (eGFR <15), but not on dialysis. They will have body composition measured, and eGFR measured.
  Interventions: Diagnostic Test: Cystatin C eGFR; Other: Bioimpedance Analysis (Body composition analysis)

INTERVENTIONS:
Diagnostic Test: Cystatin C eGFR — Cystatin C eGFR is not used routinely currently in clinical practice in the UK. It involved a blood test to analyse Cystatin C.
Other: Bioimpedance Analysis (Body composition analysis) — Participants will stand on a bioimpedance analysis machine which will measure different components of body composition

SUMMARY:
The aim of this research study is to look at the body composition (such as muscle and fat) in people with chronic kidney disease (CKD) and comparing it with body composition is people without CKD. The investigators currently understand loss of muscle function and mass (sarcopenia) affect the general health of people as they age, but this process seems to be more common, accelerated, and occurs earlier in people with CKD. There is limited evidence in this area, and we believe that if we understand when and how sarcopenia affects people with CKD, investigators can guide future trials and treatments to help treat sarcopenia, and in turn improve quality of life and health outcomes in people with CKD.

DETAILED DESCRIPTION:
In this study, the investigators will follow up people with CKD in two visits a year apart. In both visits, the investigators will measure the participants body composition and estimated kidney function using 2 different testing methods - Cystatin C eGFR and Creatinine eGFR. Using both the results in a formula, the creatinine muscle index can be calculated. If this index correlated with sarcopenia, it will be helpful tool in the care of people with CKD as will be a easy to use screening tool for sarcopenia in this population.

ELIGIBILITY:
Inclusion Criteria:

Subjects capable of giving informed consent

≥18 years of age Chronic kidney disease stages 3-5 looked after in secondary care nephrology Healthy volunteers with normal kidney function (Control)

Exclusion Criteria:

* Pregnancy
* Subjects with known neuromuscular diseases, e.g. myopathy, muscular dystrophy, muscular atrophy
* Renal transplant recipients
* Patients with pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 participants with different levels of renal function (normal renal function, CKD3,4 and 5) to be recruited from secondary care renal department.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Creatinine Muscle Index (mg/day per 1.73m2) | Day 1 (day recruited) and at 1 year
  Product of serum Creatinine and estimated glomerular filtration rate with Cystatin C (eGFRcys)

SECONDARY OUTCOMES:
Skeletal muscle mass (kg) | At Day 1 (day recruited) and 1 year
  Measured by Bioimpedance analysis
Multimorbidity Score | Day 1 (day recruited) and 1 year
  The Cambridge Multimorbidity Score is a UK validated index to score the comorbidities of participants. One can score from 0 to 20 on this index. Higher scores are associated with worse clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby and Burton NHS Foundation Trust, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No